CLINICAL TRIAL: NCT00575406
Title: Multicentre Study to Determine the Cardiotoxicity of R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristin and Prednisolone) Compared to R-COMP (Rituximab, Cyclophosphamide, Liposomal Doxorubicin, Vincristin and Prednisolone) in Patients With Diffuse Large B-Cell Lymphoma (NHL-14)
Brief Title: Multicentre Study to Determine the Cardiotoxicity of R-CHOP Compared to R-COMP in Patients With Diffuse Large B-Cell Lymphoma
Acronym: NHL-14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL-14; EudraCT 2007-004970-24
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; liposomal doxorubicin; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-CHOP (Active Comparator): Treatment with Rituximab, Cyclophosphamide, Doxorubicin, Vincristin and Prednisolone
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristin; Drug: Prednisolone
- R-COMP (Experimental): Treatment with Rituximab, Cyclophosphamide, liposomal Doxorubicin, Vincristin and Prednisolone
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: liposomal Doxorubicin; Drug: Vincristin; Drug: Prednisolone

INTERVENTIONS:
Drug: Rituximab — i.v., 375 mg/m2, d0 or d1 of each treatment cycle
  Other Names: MabThera
Drug: Cyclophosphamide — i.v., 750 mg/m2, d1 of each treatment cycle
  Other Names: Cytoxan
Drug: Doxorubicin — i.v., 50 mg/m2, d1 of each treatment cycle
  Other Names: Adriamycin
  Arms: R-CHOP
Drug: liposomal Doxorubicin — i.v., 50 mg/m2, d1 of each treatment cycle
  Other Names: Myocet
  Arms: R-COMP
Drug: Vincristin — i.v., 2mg, d1 of each treatment cycle
  Other Names: Oncovin
Drug: Prednisolone — p.o., 100mg, d1 - d5 of each treatment cycle

SUMMARY:
Diffuse large B-cell lymphoma is the most prevalent subgroup within malignant lymphoma. Clinical benefit has been shown for the treatment with cyclophosphamide, doxorubicin, vincristin and prednisolone (CHOP regimen); this could be further improved recently by the addition of rituximab (R-CHOP), a monoclonal antibody.

Improved response and overall survival rates make it necessary to evaluate late toxicities of the therapy regimens. Cardiotoxicity is a known risk factor of specific chemotherapies, with 7% patients being affected if doxorubicin cumulative doses are under 550mg/sqm. Retrospective data analyses indicate that this incidence of cardiotoxicity may be higher under combination chemotherapy. Liposomal doxorubicin has been shown to have lower cardiotoxic effects and at the same time equivalent or higher efficacy compared to conventional doxorubicin.

The aim of this study is to evaluate alternative regimens for the treatment of diffuse large B-cell lymphoma, substituting liposomal doxorubicin (R-COMP) for conventional doxorubicin (R-CHOP).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, CD20 positive, diffuse large B-cell lymphoma (DLCL)
* measurable disease according to international criteria
* male or female
* age 18 years and above
* written informed consent

Exclusion Criteria:

* myocardial infarction within 6 months prior to study entry
* cardiac insufficiency NYHA grade 3 or 4
* previous treatment with chemotherapy or radiotherapy
* CNS involvement of the disease
* positive for HIV
* WHO Performance Index 3 or 4
* secondary malignoma
* concurrent disease that prohibits chemotherapy
* known hypersensitivity towards the study interventions or their constituents
* neutropenia or thrombopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Reduction of cardiotoxicity in the R-COMP arm versus R-CHOP | Study duration

SECONDARY OUTCOMES:
Significance of serial NT-proBNP measurements for determination of anthracycline-dependent cardiotoxicity | Study Duration
Feasibility of evaluation with Haematopoietic Cell Transplantation Comorbidity Index (HCT-CI) | Study duration
Rate of Complete Responses | At end of treatment
Difference in Overall Survival at 3 and 5 yrs | 5 years
Difference in Event-free Survival at 3 and 5 yrs | 5 years
Difference in Progression-free Survival at 3 and 5 yrs | 5 years
Difference in cause-specific death | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Fridrik, MD, Principal Investigator — AKh Linz
Locations (10):
- Austria (10):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Universitaetsklinik Innsbruck/ Klinik für Innere Medizin, Innsbruck
  - A.ö. Landeskrankenhaus Leoben, Leoben
  - Krankenhaus d. Barmherzigen Schwestern Linz, Linz
  - Krankenhaus der Elisabethinen Linz, Linz
  - Krankenhaus der Stadt Linz, Linz
  - Universitaetsklinik f. Innere Medizin III, Salzburg
  - AKH Wien / Haematologie u. Haemostaseologie, Vienna
  - Hanusch Krankenhaus, Vienna
  - Klinikum Kreuzschwestern Wels GmbH, Wels